CLINICAL TRIAL: NCT03160781
Title: Pilot Study to Evaluate Combination of Intraosseous With Intra-articular Infiltrations of Plasma Rich in Growth Factors (PRGF®-Endoret®) in the Treatment of Knee Osteoarthritis.
Brief Title: Intraosseous PRP for Knee Osteoarthritis: Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unidad de Cirugía Artroscópica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCA-01-EC/13/ART
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Platelet Rich Plasma (Experimental): Combination of Intraarticular and Intraosseous Administraion of Platelet Rich Plasma
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Platelet Rich Plasma — Combination of Intraosseous and Intraarticular Infiltration of Platelet Rich Plasma

SUMMARY:
The aim of this study was to assess a novel approach to treating severe knee osteoarthritis by targeting synovialmembrane, superficial articular cartilage, synovial fluid, and subchondral bone by combining intra-articular injections and intraosseous infiltrations of platelet rich plasma.This study explored a new strategy consisting of intraosseous infiltrations of platelet rich plasma into the subchondral bone in combination with the conventional intra-articular injection in order to tackle several knee joint tissues simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 40 to 77 years.
* Predominant internal tibiofemoral knee osteoarthritis.
* Joint pain above 2.5 VAS points.
* Radiographic severity degrees 3 and 4 according to Ahlbäck scale.
* Values of body mass index between 20 and 33.
* Possibility for observation during the follow-up period.

Exclusion Criteria:

* Bilateral knee osteoarthritis which requires infiltration in both knees.
* Values of body mass index > 33.
* Polyarticular disease diagnosed.
* Severe mechanical deformity (diaphyseal varus of 4∘ and valgus of 16∘).
* Arthroscopy in the last year prior to treatment.
* Intra-articular infiltration of hyaluronic acid in the past 6 months.
* Systemic autoimmune rheumatic disease (connective tissue diseases and systemic necrotizing vasculitis).
* Poorly controlled diabetes mellitus (glycosylated hemoglobin above 9%).
* Blood disorders (thrombopathy, thrombocytopenia, and anemia with Hb < 9).
* Undergoing immunosuppressive therapy and/or warfarin.
* Treatment with corticosteroids during the 6 months prior to inclusion in the study.

Ages: 40 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2015-01-10 (Actual); Study Completion 2015-01-10 (Actual)

PRIMARY OUTCOMES:
Pain according to KOOS scale at 6 months after treatment | 6 months
  Pain according to KOOS scale

SECONDARY OUTCOMES:
Symptoms according to KOOS scale at 6 months after treatment | 6 months
  According to KOOS scale
Function according to KOOS scale at 6 months after treatment | 6 months
  According to KOOS scale
Sport Activity according to KOOS scale at 6 months after treatment | 6 months
  According to KOOS scale
QoL according to KOOS scale at 6 months after treatment | 6 months
  According to KOOS scale

IPD SHARING:
Plan to Share IPD: No